CLINICAL TRIAL: NCT02579070
Title: Efficacy and Safety of Diabetic Foot Ulcer Prevention System (DFUPS) - a Single Blind Randomised Clinical Trial in Diabetic Foot Patients at High Risk of Foot Ulceration
Brief Title: Diabetic Foot Ulcer Prevention System (DFUPS) - Part 2
Acronym: DFUPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: Freeman Health System (Other); Pennine Acute Hospitals NHS Trust (Other); National Physical Laboratory (Other); University of South Wales (Other); Photometrix (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: version 1 05/10/2015
Record Dates: First submitted 2015-10-15; First posted 2015-10-19 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Diabetic Foot
Keywords: Diabetic Foot; foot temperature; diabetic foot ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- DFUPS (visual and thermal images) (Experimental): Visual and thermal imaging with DFUPS and standard foot care. The study investigator will have access to the thermal and visual images captured with DFUPS.
  Interventions: Device: DFUPS
- DFUPS ( visual images) (Placebo Comparator): Visual and blinded thermal imaging with DFUPS and standard foot care. The study investigator will have access only to the visual images and will be blinded to the thermal images which will be captured at each visit but accessed only at the end of the study.
  Interventions: Device: DFUPS

INTERVENTIONS:
Device: DFUPS — The DFUPS device is a two-camera instrument for capturing images of feet.

SUMMARY:
The purpose of this study is to investigate whether regular measurement of skin foot temperature with a novel device (DFUPS) will prevent ulcer recurrence in diabetic patients at high risk of foot ulceration. It is planned to regularly measure the temperature of the feet of people with diabetes who have already had a foot ulcer which has subsequently healed. These measurements should allow the identification of hotspots on the foot and may be helpful when advising about ulcer risk and providing preventative treatment. It is hoped to find out whether the regular use of thermal images taken with the DFUPS device together with standard foot treatment may reduce the number of people with diabetes developing ulcers or even prevent foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Has either type 1 or type 2 diabetes
* Has intact feet as defined by the absence of a skin breakdown below the malleoli.
* Has neuropathy confirmed by impaired sensation to neurothesiometer (vibration perception threshold > 25 volts on one OR both feet)
* Has a past history of ≥1 foot ulceration (s) which has (have) resolved in the last 3 months
* Has palpable foot pulses on both feet (palpable posterior tibial artery pulse OR dorsalis pedis artery pulse OR both)
* Has no history of peripheral arterial disease
* Has footwear which in the opinion of the investigator is not likely to cause pressure damage
* Must be able to provide meaningful written informed consent for the study

Exclusion Criteria:

* Is aged <18
* Has foot deformity that in the opinion of the investigator would interfere with the interpreting of the results of the study.
* Has previous history of foot surgery which in the opinion of the study investigator could interfere with the interpreting the results of the study
* Has active foot ulceration and infection
* Has active Charcot osteoarthropathy
* Has established Charcot foot deformity that in the opinion of the study investigator would interfere with the interpreting of the results of the study.
* Has any uncontrolled illness that, in the opinion of the study investigator, would interfere with interpreting the results of the study
* Has an implantable electronic device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-02-08 (Actual); Primary Completion 2017-09-27 (Actual); Study Completion 2017-09-27 (Actual)

PRIMARY OUTCOMES:
Percentage of patients developing a foot ulcer | 12 months

SECONDARY OUTCOMES:
Time to ulceration | 12 months
Rate of change of score in quality of life from baseline and up to the final visit using the EQ-5D-5L | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Edmonds, MD, FRCP, Principal Investigator — King's College Hospital NHS Trust
Locations (3):
- United Kingdom (3):
  - King's College Hospital, London
  - The Pennine Acute Hospitals NHS Trust, Manchester
  - The Newcastle upon Tyne Hospitals, Newcastle upon Tyne